CLINICAL TRIAL: NCT05816707
Title: The Assessment of Curcuma Longa Potentials for Soft and Hard Tissue Healing in Fresh Extraction Sockets; Randomized Controlled Clinical Trial.
Brief Title: The Assessment of Curcuma Longa Potentials for Soft and Hard Tissue Healing in Fresh
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rania Farouk Mohamed Abdulmaguid (Other)
Responsible Party: Sponsor-Investigator, Rania Farouk Mohamed Abdulmaguid, Associate Professor Oral medicine and periodontology faculty of dentistry MSA university, October University for Modern Sciences and Arts
Organization: October University for Modern Sciences and Arts (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC-D652-3
Record Dates: First submitted 2023-03-19; First posted 2023-04-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Tooth Extraction Status Nos; Tooth Fracture
MeSH Terms: conditions — Tooth Fractures

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): extraction socket .
  Interventions: Other: extraction socket
- PRF Group (Active Comparator): extraction socket and PRF
  Interventions: Biological: PRF; Other: extraction socket
- Curcuma Longa Group (Active Comparator): Extraction Socket and Curcuma Longa
  Interventions: Biological: Curcuma Longa gel; Other: extraction socket

INTERVENTIONS:
Biological: PRF — Teeth will be extracted a-traumatically as possible to avoid any soft tissue or bony damage.
  The extracted sockets will be debrided by bone curettes and saline. The three extraction sockets will be divided into three groups: control group, curcumin group, and PRF group.
  After curcumin/ PRF placement, all sockets will be closed by simple interrupted suture
  Arms: PRF Group
Biological: Curcuma Longa gel — Curcuma Longa gel
  Arms: Curcuma Longa Group
Other: extraction socket — extraction socket

SUMMARY:
The study will be conducted on 30 patients with split mouth design patients will be divided into curcumin and PRF groups patients will have bilateral tooth extraction one side will receive curcumin/PRF and the other side will be control soft tissue healing and bone quality will be evaluated post-operative

DETAILED DESCRIPTION:
30 Patients will be collected from the outpatient clinic of the Department of Oral &Maxillofacial surgery, Faculty of Dentistry, MSA University, Cairo, Egypt

Eligibility criteria:

Inclusion Criteria for participants:

1. Patients with bilateral badly decayed mandibular posterior tooth that need extraction.
2. Patients free from any systemic disease
3. Patients who approved to be included in the trial and signed the informed consent.
4. Patients with no signs or symptoms of acute periapical\ periodontal infection.
5. Adults aged between 18-50 years old.

Exclusion criteria for participants:

1. Patients who are allergic to Curcumin
2. Smoker patient
3. Patients receiving chemotherapy or radiotherapy.
4. Patients who refused to be included in the trial.

Interventions:

1. Diagnosis

   * All patients will be diagnosed and selected according to inclusion and exclusion criteria.
   * Comprehensive clinical examination and understanding of patient's chief complains and needs will be done.
   * Standard preoperative intra-oral photographs (occlusal and lateral)
   * (Pre-operative orthopantogram* will be taken to ensure absence of any periapical infection)
2. Intra-operative procedures:

   Local anesthesia* will be injected intraoral around selected teeth. Patients will rinse by antiseptic mouthwash** 30 seconds before extraction. Teeth will be extracted a-traumatically as possible to avoid any soft tissue or bony damage.

   The extracted sockets will be debrided by bone curettes and saline. The three extraction sockets will be divided into three groups: control group, curcumin group, and PRF group.

   After curcumin/ PRF placement, all sockets will be closed by simple interrupted suture***
3. Postoperative treatment Analgesics **** every 6 hours for 3 days
4. Concomitant care None needed.
5. Follow up & Evaluation.

   * The extraction site will be inspected clinically after 3 days for signs of infection.
   * Soft tissue healing and pain score will be assessed after 7, 14, and 21 days.
   * 3 months post-operatively, each patient will undergo radiographic assessment by using Cone Beam Computed Tomography****** (CBCT) to evaluate bone healing and bone density.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with bilateral badly decayed mandibular posterior tooth that need extraction.

  2. Patients free from any systemic disease 3. Patients who approved to be included in the trial and signed the informed consent.

  4. Patients with no signs or symptoms of acute periapical\ periodontal infection.

  5. Adults aged between 18-50 years old.

Exclusion Criteria:

* 1. Patients who are allergic to Curcumin 2. Smoker patient 3. Patients receiving chemotherapy or radiotherapy. 4. Patients who refused to be included in the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Soft tissue healing | 21 days after surgery
  Healing index (change is being assessed)

SECONDARY OUTCOMES:
Bone Density | 3 months after surgery
  CBCT (change is being assessed)

CONTACTS AND LOCATIONS:
Locations (1):
- Rania Farouk, Cairo, Egypt